CLINICAL TRIAL: NCT06606639
Title: Reproducibility of the Acute Effect of Caffeine on Energy Metabolism and Muscular Strength, Power and Endurance Performance
Brief Title: Reproducibility of Acute Caffeine Effect
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alcala (Other)
Responsible Party: Principal Investigator, Alberto Pérez-López, Principal Investigator, University of Alcala
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Other
Other Study IDs: CEID/2024/2/039
Record Dates: First submitted 2024-09-09; First posted 2024-09-23 (Actual); Last update posted 2025-05-25 (Actual); Status verified 2025-05

CONDITIONS: Caffeine and Resistance Exercise
MeSH Terms: interventions — Caffeine

STUDY DESIGN:
Who Masked: Participant, Investigator
Masking Description: Statistician
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (5):
- Caffeine - Trial 1 (Experimental)
  Interventions: Dietary Supplement: Caffeine
- Caffeine - Trial 2 (Experimental)
  Interventions: Dietary Supplement: Caffeine
- Caffeine - Trial 3 (Experimental)
  Interventions: Dietary Supplement: Caffeine
- Placebo - Trial 1 (Placebo Comparator)
  Interventions: Dietary Supplement: Placebo
- Placebo - Trial 2 (Placebo Comparator)
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Caffeine — acute caffeine intake (3 mg/kg)
  Arms: Caffeine - Trial 1; Caffeine - Trial 2; Caffeine - Trial 3
Dietary Supplement: Placebo — Acute placebo intake (3 mg/kg of maltodextrin)
  Arms: Placebo - Trial 1; Placebo - Trial 2

SUMMARY:
Introduction: Various studies have evaluated and verified the ergogenic effect of acute caffeine intake on sports performance, specifically on strength and power performance. However, all experimental investigations designed so far have been based on the comparison of the "caffeine" and "placebo" conditions in a single trial, not considering the reproducibility and variability of caffeine in multiple trials.

Objectives: The present study aims to evaluate the reproducibility and replicability of the acute effect of caffeine intake on energy metabolism and the muscular production of force, power and endurance, according to sex (men vs women) and type of exercise ( bench press vs squat).

ELIGIBILITY:
Inclusion Criteria:

* Age between ≥ 18 and ≤ 35 years.
* Body Mass Index (BMI) < 25 kg/m².
* Resistance-trained individuals (> 2 years of structured trained).
* Healthy men and women without neurological, cardiometabolic, immunological, or physical conditions that prevent them from exercising.
* Participants must be able to perform the tests described in the following section.

Exclusion Criteria:

* History of neuromuscular diseases, heart diseases, or diseases that may affect liver or muscle metabolism.
* Use of drugs, other stimulants or sport supplements that interfere with the the study dietary supplement.
* Sedentary habits (<150 min/week of moderate exercise).
* Having undergone prolonged periods of forced physical inactivity during the 6 months prior to the study.
* Performing strenuous exercise during the 48 hours prior to the tests.
* Failure to replicate the same food intake on the two days of the experiments.
* Consuming caffeine or any other stimulant after 6 pm the day before the training or tests, to avoid headaches, discomfort, or lethargy among regular caffeine consumers.

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 48 (Actual)
Dates: Start 2024-01-08 (Actual); Primary Completion 2024-05-22 (Actual); Study Completion 2024-05-22 (Actual)

PRIMARY OUTCOMES:
Mean velocity at different %1RM | Through study completion, an average of 4 weeks
  Measuring bar mean velocity desplacement during bench press and back squat exercises.
Peak velocity at different %1RM | Through study completion, an average of 4 weeks
  Measuring bar peak velocity and time to reach peak velocity of bar desplacement during bench press and back squat exercises.
Mean power output at different %1RM | Through study completion, an average of 4 weeks
  Measuring during bench press and back squat exercises.
Peak power output and time to reach peak power output at different %1RM | Through study completion, an average of 4 weeks
  Measuring during bench press and back squat exercises.
Number of repetitions performed in 1 set at 65%1RM until task failure | Through study completion, an average of 4 weeks
  In bench press and back squat exercises
Bar velocity deplacement performed in 1 set at 65%1RM until task failure | Through study completion, an average of 4 weeks
  In bench press and back squat exercises
Power output generated in 1 set at 65%1RM until task failure | Through study completion, an average of 4 weeks
  In bench press and back squat exercise
Resting Metabolic Rate (RMR) | Through study completion, an average of 4 weeks
  Kcal at rest measuring (RMR) using a metabolic chart.
Maximal Fat Oxidation Rate (MFO) | Through study completion, an average of 4 weeks
  g/min (MFO) using a metabolic chart.

SECONDARY OUTCOMES:
Physical activity (METs-min/wk) | Through study completion, an average of 4 weeks
  Using IPAQ
Dietary (g/kg of macronutrients) | Through study completion, an average of 4 weeks
  Using 24-total recall
Mood state | Through study completion, an average of 4 weeks
  Mood. Participants graded a set of 29 items related to the mood on a Likert scale from 0 (not at all) to 4 (extremely) in reply to the question;How do you feel at this moment?; to assess six scales: tension, depression, anger, vigor, fatigue and confusion.
Adverse effects | Through study completion, an average of 4 weeks
  Adverse effects. perception of power, endurance, energy and exertion, as well as heart, muscular and gastrointestinal discomfort.
Fat mass | Through study completion, an average of 4 weeks
  Using electrical bioimpedance (kg and % of body mass)
Fat-free mass | Through study completion, an average of 4 weeks
  Using electrical bioimpedance (kg and % of body mass)

CONTACTS AND LOCATIONS:
Locations (1):
- Facultad de Medicina y Ciencias de la Salud. Universidad de Alcalá, Alcalá de Henares, Madrid, Spain

IPD SHARING:
Plan to Share IPD: Yes